

#### STATISTICAL ANALYSIS PLAN

**Study Title:** An Extension Study to Investigate the Safety and Durability of

Clinical Activity of Idelalisib in Subjects with Hematologic

Malignancies

Name of Test Drug: Idelalisib (IDELA; GS-1101)

Study Number: 101-99

**Protocol Version:** Amendment 1

**Protocol Date:** 12 April 2010

**Analysis Type:** End of Study

**Analysis Plan Version:** Version 1.0

Analysis Plan Date: 01 April 2013

Analysis Plan Author: PPD

## CONFIDENTIAL AND PROPRIETARY INFORMATION

## **TABLE OF CONTENTS**

| TAB | SLE OF | CONTENTS | 2 |
|---|---|---|---|
| LIST | OF IN | -TEXT TABLES | 3 |
| LIST | OF A | BBREVIATIONS | 4 |
| 1. | INTRO | DDUCTION | 5 |
| 1. | 1.1. | Study Objectives | |
| | 1.1. | Study Objectives | |
| | 1.3. | Sample Size and Power | |
| 2. | ТҮРЕ | OF PLANNED ANALYSIS | |
| 3. | GENE | RAL CONSIDERATIONS FOR DATA ANALYSES | 12 |
| | 3.1. | Analysis Sets | 12 |
| | | 3.1.1. Intent-to-Treat Analysis Set | 12 |
| | 3.2. | Subject Groups | |
| | 3.3. | Treatment Strata | 12 |
| | 3.4. | Examination of Subject Subsets | |
| | 3.5. | Multiple Comparisons. | |
| | 3.6. | Missing Data and Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | |
| | 2.0 | 3.7.1. Data Handling for Efficacy Endpoints | |
| | 3.8. | Visit Windows | |
| | | 3.8.1. Definition of Study Day 1 and Baseline | |
| | | 3.8.3. Selection of Data in the Event of Multiple Records in a Window | |
| 4. | SUBJI | ECT DISPOSITION | |
| | 4.1.<br>4.2. | Disposition of Subjects | |
| | 4.2. | 4.2.1. Duration of Exposure to Study Drug | |
| | 4.3. | Protocol Deviations | |
| 5. | | LINE DATA | |
| | 5.1. | Demographics and Baseline Characteristics | |
| | 5.1. | Disease History | |
| | 5.3. | Medical History | |
| | | • | |
| 6. | | ACY ANALYSES | |
| | 6.1. | Definition of the Efficacy Endpoints | 19 |
| | | 6.1.1. Overall Response Rate (ORR) | |
| | | 6.1.2. Duration of Response (DOR) | |
| | | 6.1.3. Progression-Free survival (PFS) | |
| | 6.2. | 6.1.4. Time to Response (TTR) | |
| | 6.3. | Analysis of the Efficacy Endpoint | |
| | 0.5. | 6.3.1. Overall Response Rate (ORR) | |
| | | 6.3.2. Time-to-Event Endpoints | |
| | | 6.3.3. Time to Response (TTR) | |
| | | 6.3.4. Sensitivity Analysis | |
| | 6.4. | Changes From Protocol-Specified Efficacy Analyses | |

| 7. | SAFE | ETY ANALYSES | 22 |
|---|---|---|---|
| | 7.1. | Adverse Events and Deaths | 22 |
| | | 7.1.1. Adverse Event Dictionary | |
| | | 7.1.2. Adverse Event Severity | |
| | | 7.1.3. Relationship of Adverse Events to Study Dru | |
| | | 7.1.4. Serious Adverse Events | |
| | | 7.1.5. Treatment-Emergent Adverse Events | 24 |
| | | 7.1.5.1. Definition of Treatment-Emerg | ent24 |
| | | 7.1.5.2. Incomplete Dates | 24 |
| | | 7.1.6. Summaries of Adverse Events and Deaths | 24 |
| | 7.2. | Allowed Concomitant Therapy | 20 |
| | 7.3. | Prior Therapy | 20 |
| | 7.4. | Physical Examination | 20 |
| | 7.5. Changes From Protocol-Specified Safety Analyses | | |
| 8. | SOFT | ΓWARE | 28 |
| 9. | SAP F | REVISION | 29 |
| 10. | APPE | ENDICES | 30 |
| | 10.1. | Tables | 30 |
| | 10.2. | Listings | 7: |
| | 10.3. | Figures | 7 <sup>′</sup> |
| | | LIST OF IN-TEXT TAB | LES |
| | Table | e 1. Overview of Clinical Studies | |

#### LIST OF ABBREVIATIONS

AE adverse event BID twice a day

CI confidence interval

CLL chronic lymphocytic leukemia

CR complete response
CRF case report form
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

CYP cytochrome P450

DLBCL diffuse large B-cell lymphoma FDA Food and Drug Administration

FL follicular lymphoma
HLGT high-level group term
HLT high-level term

ICH International Conference on Harmonisation

iNHL indolent non-Hodgkin lymphoma

LLT low level term

LPL/WM lymphoplasmacytic lymphoma/ Waldenström's macroglobulinemia

MCL mantle cell lymphoma

MedDRA Medical Dictionary for Regulatory Activities

MR minor response

NHL non-Hodgkin lymphoma PD progressive disease

PI3K phosphatidylinositol 3-kinase PFS progression-free survival

PR partial response
PT preferred term
Q1 quartile 1
Q3 quartile 3

SAE serious adverse event SAP statistical analysis plan

SD stable disease SE standard error

SLL small lymphocytic lymphoma

SOC system organ class StD standard deviation

TEAE treatment-emergent adverse event
TFLs tables, figures, and listings
WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

WM Waldenström's macroglobulinemia

### 1. INTRODUCTION

Study 101-99 is an extension study which provides the opportunity for subjects with hematologic malignancies who complete a prior idelalisib (IDELA) study protocol (including Studies 101-02, 101-07, 101-08 and 101-10) to continue IDELA treatment as long as the subject is deriving clinical benefit.

Study 101-02 was a Phase 1 monotherapy study in subjects with selected, relapsed, or refractory hematologic malignancies. This study was the first in which IDELA was administered to subjects with hematologic malignancies. Its objective was to collect initial IDELA safety and pharmacology data to identify dosing regimens for subsequent clinical trials.

Studies 101-07 and 101-08 are both combination studies. 101-07 is a Phase 1 study to investigate the safety and clinical activity of IDELA in combination with chemotherapeutic agents and anti-CD20 mAb in subjects with relapsed or refractory indolent non-Hodgkin lymphoma (iNHL), mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL). Study 101-08 is a Phase 2 single-arm study to investigate the safety and clinical activity of IDELA in combination with rituximab in elderly subjects with previously untreated CLL or small lymphocytic lymphoma (SLL).

Study 101-10 is a Phase 1/2, uncontrolled study of IDELA in subjects with previously treated low-grade iNHL. The objective of this study is to investigate the safety and efficacy of IDELA in those subjects.

Table 1 provides an overview of each of the 4 clinical studies:

Table 1.Overview of Clinical Studies

| Study | Study Design | Diseases | Objectives | Dosage and Regimen | Status |
|---|---|---|---|---|---|
| 101-02 | Phase 1, sequential dose-<br>escalation study of<br>IDELA in subjects with<br>select, relapsed or<br>refractory hematologic<br>malignancies | Relapsed or<br>refractory CLL,<br>iNHL, MCL,<br>DLBCL, AML,<br>or MM | Safety,<br>activity, PK,<br>PD | IDELA x 28 days:<br>50, 100, 150, 200,<br>350 mg BID;<br>150, 300 mg once daily<br>up to 48 weeks<br>IDELA x 21 days/7 days<br>off:<br>150 mg BID up to<br>48 weeks | Complete |
| 101-08 | Phase 2, single-arm study<br>of IDELA in combination<br>with rituximab in elderly<br>subjects with previously<br>untreated CLL or SLL | Untreated CLL<br>or SLL | Efficacy,<br>safety, PK, PD | IDELA:<br>100 or 150 mg BID x<br>48 weeks<br>Rituximab:<br>375 mg/m <sup>2</sup> IV weekly x<br>8 weeks | Ongoing |
| 101-10 | Phase 1/2, single-agent,<br>uncontrolled study of<br>IDELA in subjects with<br>previously treated low-<br>grade (indolent) NHL | Relapsed or<br>refractory iNHL | Safety,<br>efficacy, flow<br>cytometry | IDELA 150 mg BID for<br>28-day cycles up to<br>12 cycles | Ongoing |

| Study | Study Design | Diseases | Objectives | Dosage and Regimen | Status |
|---|---|---|---|---|---|
| 101-07 | Phase 1 study of IDELA in combination with chemotherapeutic agents and anti-CD20 mAb in relapsed or refractory iNHL or CLL | Relapsed or refractory iNHL or CLL | Safety,<br>activity, PK,<br>PD | IDELA: 100 or 150 mg BID continuously up to 48 weeks given in combination with: Rituximab: 375 mg/m² IV weekly x 8 weeks Bendamustine: 70 or 90 mg/m² IV Days 1 and 2 every 4 weeks x 24 weeks Rituximab-Bendamustine Rituximab-Bendamustine Rituximab 375 mg/m² IV every 4 weeks x 24 weeks, and Bendamustine 70 or 90 mg/m² IV Days 1 and 2 every 4 weeks x 24 or 48 weeks Ofatumumab: 300 mg IV Day 1 or 2, then 1000 mg weekly for Weeks 2-8, followed by 1000 mg every 4 weeks for 4 doses during Weeks 9-12 Fludarabine: 40 mg/m² PO Days 1-5 every 4 weeks x 24 weeks Everolimus: 10 mg PO Days 1-28 of every 4-week cycle Bortezomib: 1.3 mg/m² SC Days 1, 8, and 15 every 4 weeks Chlorambucil: 10 mg/m² PO Days 1-7 every 4 weeks x 48 weeks | Ongoing |

The purpose of this statistical analysis plan (SAP) is to provide a framework based on which the protocol objectives may be achieved in a statistically rigorous fashion, with minimal bias or analytical deficiencies. Specifically, this SAP is intended to prospectively (a priori) outline

the types of data analyses that will attempt to answer the study objectives outlined in the protocol. The plan explains the data-handling methods and analyses and adheres to commonly accepted practices of biostatistical analysis in the pharmaceutical industry.

The analyses outlined in this plan are based upon the protocol for Study 101-99.

## 1.1. Study Objectives

| Primary Study Objectives | To investigate the long-term safety of IDELA in subjects with hematologic malignancies |
|---|---|
| | To determine the duration of clinical benefit of IDELA in subjects with hematologic malignancies |
| <b>Secondary Study Objectives</b> | There are no secondary objectives for this study. |

## 1.2. Study Design

| Design Configuration and Subject Population | Subjects with hematologic malignancies completing a prior IDELA study with a clinical benefit are eligible for enrollment in the study. Subjects will be followed according to the standard of care as appropriate for the underlining disease. |
|---|---|
| | Subjects entered into the study will have one of the following diagnoses: |
| | • CLL |
| | • Indolent B-cell NHL (iNHL) |
| | Small lymphocytic lymphoma (SLL) |
| | Lymphoplasmacytic<br>lymphoma/Waldenstrom's<br>macroglobulinemia (LPL/WM) |
| | Splenic marginal zone lymphoma |
| | • Follicular lymphoma (FL) |
| | Extranodal marginal zone B-cell lymphoma |
| | Nodal marginal zone B-cell lymphoma |
| | Aggressive B-cell NHL |
| | Mantle cell lymphoma (MCL) |
| | Diffuse large B-cell lymphoma (DLBCL) |

| Treatment Groups | The dose of IDELA will generally be the same as the dose that was administered at the end of the prior study. Subjects will not be randomized to a different dose. |
|---|---|
| Study Periods/Phases | After entering the study, subjects will continue to receive treatment as long as they are deriving clinical benefit. A subject may be withdrawn from the study under the following circumstances: |
| | The subject wishes to withdraw consent to participate in the study |
| | The subject wishes to discontinue study drug treatment fro any reason |
| | The subject experiences a toxicity that necessitates discontinuing study drug treatment permanently |
| | The subject has progressive disease or is no longer deriving clinical benefit |
| | The investigator or sponsor decides to discontinue treatment for medical reasons or due to the subject's noncompliance with the protocol |
| | The Sponsor discontinues the study |
| | While on study, the subject will return every 2-months for the following procedures: |
| | Recording of grade 3 or higher adverse events<br>(AEs), all SAE and antitumor concomitant<br>medications |
| | • Return of used drug supply and dispensing of 2-months of new drug supply |
| | Subjects will also be followed for disease status according to standard of care. Any change in the clinical response status should be recorded. |

## **Schedule of Assessments**

| Randomization | No randomization or blinding will be performed in this study. |
|---|---|
| Site and/or Stratum Enrollment<br>Limits | This is a multi-center study. Data will be aggregated across all centers for analyses. Individual subject listings will identify each subject by study center. |
| Study Duration | All subjects may receive study drug indefinitely unless a withdrawal criterion is met: subjects will be withdrawn from this study if they develop progressive disease, unacceptable toxicity related to IDELA, or if they no longer derive clinical benefit in the opinion of the investigator. |

# 1.3. Sample Size and Power

| Planned Sample Size | The sample size for this study depends on the number of eligible subjects from prior studies conducted with IDELA (101-02, 101-07, 101-08 and 101-10). As such, no formal calculation is applicable. |
|---|---|
| Power Statement | Not applicable at this point in the study |
| Actual Enrollment and Impact on Power | Not applicable at this point in the study |

## 2. TYPE OF PLANNED ANALYSIS

The final analysis will be performed when all enrolled subjects have completed efficacy and safety assessments.

### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

## 3.1. Analysis Sets

#### 3.1.1. Intent-to-Treat Analysis Set

The intent-to-treat (ITT) analysis set will consist of all enrolled subjects that received any dose of IDELA in this study.

#### 3.2. Subject Groups

Study 101-99 is an extension study, therefore subject groups will follow the same categorization as the parent study for all summaries. The dose of IDELA will generally be the same as the dose that was administered at the end of the parent study.

Summary of efficacy will be presented by integrating the parent study with 101-99 for 101-02, 101-07, and 101-08, respectively. No efficacy analysis will be performed on 101-10.

Summary of safety will be presented using the following 2 data sets:

- All subjects in parent studies regardless of whether they entered 101-99, summaries will be provided combining data from both the parent study and 101-99
- Only subjects in parent studies who rolled over to 101-99
  - Summaries will be provided combining data from both the parent study and 101-99
  - Summaries will be provided only using data from 101-99

#### 3.3. Treatment Strata

Not applicable

#### 3.4. Examination of Subject Subsets

Potential subject subsets may include the following cytogenesis factors:

- 17p deletion and/or p53 mutation in CLL cells: either vs. neither
- Immunoglobulin heavy chain variable region (IgHV) mutation: unmutated vs. mutated
- Any prior therapy with an anti-CD20 therapeutic antibody: Yes vs. No

Disease history, prior therapy, and AEs will be examined depending on the following demographic characteristics:

- Sex (male vs. female)
- Age group (<65 vs>=65)
- Race (White vs. non-White)

However, the final subject categorization will depend on the actual number of subjects in each group. If there are very few subjects in the group, the subgroup analysis won't be performed.

### 3.5. Multiple Comparisons

Not applicable

#### 3.6. Missing Data and Outliers

#### **Missing Data**

A missing data point for a given study visit may be due to any of the following reasons:

- A visit occurred in the window but data were not collected or were unusable
- A visit did not occur in the window
- A subject permanently discontinued from the study before reaching the window.

Analyses will be based upon observed data without imputation.

#### **Outliers**

Outliers won't be excluded unless otherwise specified.

### 3.7. Data Handling Conventions and Transformations

- By-subject listings will be presented for subjects in the ITT analysis set and sorted by subject number, visit, and time (if applicable).
- Summary tables for continuous variables will contain the following statistics: N (number in analysis set), n (number with data), mean, standard deviation (STD), 95% CI, median, Q1, Q3, minimum, and maximum. The same number of decimal places as in the raw data will be presented when reporting minimum and maximum, 1 more decimal place than in the raw data will be presented when reporting mean, median, Q1 and Q3, and 2 more decimal places than in the raw data will be presented when reporting STD and 95% CI.

- Summary tables for categorical variables for baseline and safety data will include: N, n, percentage. The tables for efficacy endpoints will include standard error, and 95% CIs on the percentage, where appropriate. Unless otherwise indicated, 95% CIs for binary variables will be calculated using the binomial distribution. The denominator for the percentages will be the number of subjects in the respective analysis set, unless otherwise specified. Missing data will be included as a row in tables where it is appropriate. All percentages will be presented as one-decimal point, unless otherwise specified. Percents equal to 100 will be presented as 100% and percents will not be presented for zero frequencies.
- Unless otherwise specified, all analyses will be 2-sided at the 0.05 level of significance. P-values should be rounded to 3 decimal places. Any p-value less than 0.001 will be presented as < 0.001.
- For Kaplan-Meier (KM) estimates, the 95% CIs will be calculated using the Greenwood's formula with (complementary) log-log transformation.
- Unscheduled visits will be only included in listings and the best or worst post-baseline summary. Unscheduled visits will not be included in the by-visit summary tables, unless otherwise specified.

All displays will be produced using the Times New Roman font size 9.

#### 3.7.1. Data Handling for Efficacy Endpoints

If there is a significant degree of non-normality for a continuous endpoint, analysis may be performed on log-transformed data or nonparametric method, as appropriate.

#### 3.8. Visit Windows

### 3.8.1. Definition of Study Day 1 and Baseline

Study Day 1 is defined as the day of first dose of study drug from the parent study.

Baseline is defined as the last observation before the first dose from the parent study unless otherwise specified.

#### 3.8.2. Analysis Windows

For parameters that will be summarized by visit, the nominal visit as recorded on the electronic case report form will be used. For parameters assessed at the end of treatment (EOT) visit, the assessment results will be assigned to the next schedule visits where the respective data were scheduled to be collected for summary. There will be no additional analysis windowing done based on the assessment date.

## 3.8.3. Selection of Data in the Event of Multiple Records in a Window

For summary purposes, when a single value at a visit is needed, the following rules will be used:

- The observation that is closest to the target visit as defined in the protocol will be used in the analyses if there are multiple observations in a visit.
- The latest one will be used if observations have the same distance (before and after) to the target visit.
- The last measurement will be used if multiple measurements are all taken on the same day.

### 4. SUBJECT DISPOSITION

## 4.1. Disposition of Subjects

The number and percentage of subjects who received study drug, completed the parent study, entered study 101-99 and discontinued from study 101-99 will be summarized. Subjects who discontinued study 101-99 for the following reasons will be summarized: AE, withdrew consent, patient request, investigator request, disease progression, death, sponsor discontinued study and other. A summary will be provided separately for each individual study with 101-99.

The disposition data will be presented in the subject data listings.

#### 4.2. Extent of Exposure

### 4.2.1. **Duration of Exposure to Study Drug**

Duration of exposure of study drug in months will be defined as (last dose date – Study Day 1 + 1) / 30.4375, regardless of temporary interruptions in study drug administration. For subjects who entered 101-99 and are still on study, the date of data cut-off will be used to calculate duration of exposure, (data cut-off date – Study Day 1 + 1) / 30.4375. Date of Study Day 1 will be obtained from the parent study. Duration of exposure of study drug will be summarized using descriptive statistics (n, mean, StD, median, Q1, Q3, minimum and maximum) and as the number and percentage of subjects categorized by exposure at least 1 day, 2, 4, 6, 12, 18, 24, 30, and 36 months, respectively.

#### 4.3. Protocol Deviations

Protocol deviations will be identified before database lock by the Gilead clinical team. Important (major) protocol deviations will be summarized by type of deviation in the clinical study report (CSR). A listing will be provided for all major protocol deviations.

### 5. BASELINE DATA

### 5.1. Demographics and Baseline Characteristics

Demographics and baseline characteristics information will be captured from the parent study.

Demography including gender, race, ethnicity, age (years), weight (kg), height (cm), and body mass index (BMI, kg/m²) will be summarized for the ITT Analysis Set. Gender, race, ethnicity, and WHO performance score will be summarized by using summary statistics for categorical variables. Age, weight, height, and BMI will be summarized by using summary statistics for continuous variables.

Age will be calculated as the number of years between date of birth and date of first dosing.

Age (years) = (date of first dose of study drug in the parent study – date of birth+1) / 365.25 (round down to an integer)

BMI  $(kg/m^2)$  = weight /  $(height)^2$  (round to 1 decimal point)

Summary will be provided separately for each individual study with 101-99, but will only include subjects who rolled over to 101-99.

All demographic and baseline characteristics data described above will be presented in the subject data listings.

## 5.2. Disease History

Disease history information will be captured from the parent study.

Disease history including subjects' disease stage and disease status etc will be summarized and listed separately for each individual study on subjects who entered 101-99.

Partial date of diagnosis will be imputed as follows:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month.

No imputation will be done if the year of diagnosis is missing.

## **5.3.** Medical History

Medical history information will be captured from the parent study.

For 101-02 and 101-10, medical conditions are categorized by body system. For 101-07 and 101-08, medical conditions will be coded by system organ class (SOC), high level term (HLT), and preferred term (PT) by using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary version 15.1. Ongoing medical conditions will be graded per Common Terminology Criteria for Adverse Events (CTCAE) version 4.02 (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening). Medical history data will be summarized and listed separately for each individual study based on subjects who entered 101-99.

#### 6. EFFICACY ANALYSES

The parent study will be integrated with 101-99 for efficacy analyses. The data will be summarized separately for 101-02, 101-07 and 101-08 with 101-99 based on subject disease and dose categorization as in the parent study. The analyses will be performed on all subjects enrolled in the parent study regardless of their rolling over to 101-99 or not.

#### 6.1. Definition of the Efficacy Endpoints

The efficacy endpoints include the overall response rate (ORR), duration of clinical response (DOR), progression-free survival (PFS), and time to response (TTR) based on investigator's assessment.

Response is categorized as Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD) for CLL subjects, and CR, PR, Minor Response (MR) (for LPL/WM subjects), SD, or PD for iNHL subjects.

#### 6.1.1. Overall Response Rate (ORR)

ORR is defined as the proportion of subjects who achieve a CR or PR (or MR for LPL/WM subjects) after the start of IDELA treatment until progression or the end of study drug treatment. Subjects who do not have any post baseline tumor assessments for any reason are included in the denominator when calculating the response rate based on the ITT analysis set.

#### 6.1.2. Duration of Response (DOR)

DOR is defined as the interval (in months) from the first documentation of CR or PR (or MR) to the earlier of the first documentation of disease progression or death from any cause. DOR will only be evaluated in subjects who have a response of CR or PR.

DOR = (Date of event or censoring – Date of first documentation of CR or PR (or MR) + 1) / 30.4375.

Date of first document of CR or PR (or MR) will be captured by combining the parent study with 101-99 (first response could occur in the extension study).

#### 6.1.3. Progression-Free survival (PFS)

PFS is defined as the interval (in months) from the start of IDELA treatment to the earlier of the first documentation of disease progression or death from any cause.

PFS = (Date of event or censoring – Study Day 1 + 1) / 30.4375.

Date of first documentation of CR or PR (or MR) will be captured by combining the parent study with 101-99 (first response could occur in the extension study).

#### 6.1.4. Time to Response (TTR)

TTR (months) is defined as the interval from the start of study treatment to the first documentation of CR, PR (or MR). TTR will be evaluated only for subjects who have a response of CR or PR.

TTR = (Date of first documentation of CR or PR (or MR) – Study Day 1 + 1) / 30.4375.

#### 6.2. Statistical Hypothesis for the Efficacy Endpoint

There is no formal statistical hypothesis specified for this study.

#### 6.3. Analysis of the Efficacy Endpoint

#### 6.3.1. Overall Response Rate (ORR)

The best overall response will be summarized by each response category as CR, PR, MR (for LPL/WM subjects), SD, PD, and not available (NA). The ORR will be calculated as the proportion of subjects with response (CR, PR or MR) and corresponding 2-sided 95% exact confidence interval will be provided.

Data listings for the clinical responses will be presented.

#### 6.3.2. Time-to-Event Endpoints

For time-to-event endpoints (DOR and PFS), data from surviving, non-progressing subjects will be censored at the earlier of the time of initiation of antitumor treatment other than the study treatment or at the latest time of last drug dispense and last time that lack of progression was documented.

If a subject does not have a baseline tumor assessment, then the DOR and PFS will be censored at the date of first dose of study treatment, regardless of whether or not disease progression or death has been observed.

DOR will be evaluated for subjects who achieve a response of CR, PR (or MR). DOR will also be summarized using Kaplan-Meier methods and corresponding survival curves will be plotted.

PFS will be summarized using Kaplan-Meier methods and corresponding survival curves will be plotted.

All the derived endpoints will be listed.

#### 6.3.3. Time to Response (TTR)

TTR will be evaluated for subjects who achieve a response of CR, PR (or MR). It will be summarized using descriptive statistics.

### 6.3.4. Sensitivity Analysis

Antitumor concomitant therapy is allowed in the extension study. It was used for a specific purpose, not for disease progression. Therefore the initiation of the treatment shouldn't be a sign of progression per protocol. A sensitivity analysis will be performed by not censoring DOR and PFS by subjects' use of antitumor medication in 101-99 other than the study treatment.

#### 6.4. Changes From Protocol-Specified Efficacy Analyses

The protocol specified that data will be summarized by the use or not of concomitant anti-cancer therapy. As anti-cancer therapy is allowed in this study per protocol, a summary will be given for all subjects regardless of taking antitumor treatment or not. However, a sensitivity analyses will be performed by not censoring DOR and PFS by subjects' use of anti-cancer therapy in 101-99 other than the study treatment.

ORR and TTR have been added as additional efficacy endpoints.

#### 7. SAFETY ANALYSES

The primary safety endpoint for this study will be the incidence of AEs. Only grade 3 or higher AEs and all serious adverse events (SAEs) encountered by enrolled subjects during the clinical trial from the time the informed consent for 101-99 is signed through the end of study visit are required to be recorded on the AE CRF page(s). A summary will be provided by including all AEs recorded.

The data will be summarized separately for 101-02, 101-07, 101-08 and 101-10 based on subject disease and dose categorization as in the parent study.

The summary of safety will be presented using the following 3 populations:

- Parent study integrated with 101-99: all subjects in the parent study + 101-99
- Parent study integrated with 101-99: only subjects in the parent study who rolled over to 101-99
- 101-99 alone: use data from 101-99 alone, by the parent study, including only key safety endpoints (ie, AEs Grade ≥ 3, SAEs)

No lab data are collected in 101-99 per study protocol.

#### 7.1. Adverse Events and Deaths

An AE is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. It can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical (investigational) product, whether or not related to the medicinal product. The start of the AE reporting for a study subject will coincide with signing of the informed consent. The end of the adverse-event-reporting period occurs 30 days after discontinuation from study or when any ongoing drug-related AEs and/or SAEs have resolved or become stable.

The focus of AE summarization will be on treatment-emergent AEs using the ITT analysis set. All AEs will be listed.

### 7.1.1. Adverse Event Dictionary

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 15.1). System organ class (SOC), high level group term (HLGT), high level term (HLT), preferred term (PT), and lower level term (LLT) will be attached to the clinical database.

#### 7.1.2. Adverse Event Severity

The severity of AEs will be graded by the investigator according to the CTCAE, according to the individual study protocol, whenever possible. If a CTCAE criterion does not exist, the grade corresponding to the appropriate adjective will be used by the investigator to describe the maximum intensity of the AE. The severity grade will be categorized as:

- Grade 1 (mild)
- Grade 2 (moderate)
- Grade 3 (severe)
- Grade 4 (life threatening)
- Grade 5 (fatal)

A missing severity grade will be considered as missing.

In 101-99, only grade 3 or higher AEs and all SAEs are required to be recorded on the AE CRF page(s).

#### 7.1.3. Relationship of Adverse Events to Study Drug

The investigator-described relationship of the AE to the study drug was assessed as below:

Study 101-10:

- Related
- Not related

Study 101-02, -07, -08 and -99:

- Probable
- Possible
- Unlikely
- Unrelated

AEs will be recorded as treatment-related in the CRF if the causal relationship with study drug is recorded as probable or possible. Those that are considered to be unlikely or unrelated to treatment with study drug will be recorded as not treatment-related. Events for which the investigator did not record relationship to study drug will be considered related and data listings will show relationship as missing.

#### 7.1.4. Serious Adverse Events

SAEs are those identified as serious in the clinical database. The clinical database will be reconciled with the SAE database from the Drug Safety and Public Health Department (DSPH) database finalization.

## 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment-Emergent

Treatment-emergent AEs are events in a given study period that meet one of the following criteria:

- Events with onset dates on or after the start of treatment and up to 30 days after the permanent discontinuation of the study medication.
- The continuing AEs diagnosed prior to the start of treatment and worsening in severity grade, or non-serious AEs at baseline which become serious, or AEs resulting in treatment discontinuation after the start of treatment.

#### 7.1.5.2. Incomplete Dates

All AEs with partial onset or stop dates will be identified and the partial dates will be imputed as follows:

- For AE onset date: If day and month are missing but year is available, then the imputed day and month will be 01Jan or the first dosing date if they have the same year, whichever is later. If day is missing but the month and year are available, then the imputed day will be the first day of the month or the first dosing date if they have the same month and year, whichever is later.
- For AE stop date: If day and month are missing but year is available, then the imputed day and month will be 31Dec or 30 days after the last dose of IDELA if they have the same year, whichever is earlier. If day is missing but the month and year are available, then the imputed day will be the last day of the month or 30 days after the last dose of IDELA if they have the same month and year, whichever is earlier.

#### 7.1.6. Summaries of Adverse Events and Deaths

A brief summary of treatment-emergent AEs will show the number and percentage of subjects who (1) had any AE, (2) had any Grade ≥3 AE, (3) had any treatment-related AE, (4) had any Grade ≥3 treatment-related AE, (5) had any SAE, (6) had any treatment-related SAE, (7) discontinued from study drug due to an AE, and (8) all death.

Summaries (number and percentage of subjects) of treatment-emergent AEs (by SOC, HLT and PT) will be provided as follows:

- All AEs
- All AEs by severity
- Grade  $\geq$  3 AE
- All treatment-related AEs
- Treatment-related AEs of any grade and Grade ≥3
- All SAEs
- All treatment-related SAEs
- All AEs that caused study drug dose reduction
- All AEs that caused discontinuation from study drug
- AEs leading to deaths

Multiple events will be counted once only per subject in each summary. For data presentation, SOC, HLT and PT will be sorted by decreasing frequency. For summaries by severity grade, the most severe event will be selected. In addition to the presentation by SOC and HLT, each summary listed above will also be presented by preferred term in decreasing frequency.

Summary of all treatment-emergent AEs will also be summarized by SOC, HLT and PT in the following subgroups: sex (male vs female), age group (<65 vs >=65) and race (White vs non-White) when applicable.

In addition to the by-treatment summaries, data listings will be provided for the following:

- All AEs (with a variable indicating whether the event is treatment-emergent)
- SAEs (with a variable indicating whether the event is treatment-emergent)
- AEs leading to death
- AEs leading to dose reduction of study drug
- AEs leading to discontinuation of study drug

Relative day from first dose date will be provided for each AE in the listings. If the AE onset date is after the first dose date, the relative day will be calculated as (AE onset date – first dose date + 1), however, if the AE onset date is prior to the first dose date, the relative day will be calculated as (AE onset date- first dose date).

### 7.2. Allowed Concomitant Therapy

Concomitant treatment as deemed medically necessary by the investigator is allowed in 101-99. The only antitumor therapies allowed are monoclonal antibodies for subjects with CLL who do not have an objective response to IDELA. Only anti-cancer concomitant medications will be recorded in the 101-99 CRF. A listing will be provided for all subjects taking antitumor medication in the study.

Concomitant medications will be coded using the standard World Health Organization Drug Dictionary (WHO-DD, Version 2009Q3).

### 7.3. Prior Therapy

Prior therapy information will be captured from the parent study.

Number of prior therapy regimens will be summarized using descriptive statistics. The partial completion date will be imputed using the following algorithm:

- If day and month are missing but year is available, then the imputed day and month will be 01Jan.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month.
- If year is missing, no imputation will be done and the completion date will be treated as missing.

Number of subjects who received certain regimens (eg, BR, CHOP, R-CHOP, etc.) will be summarized using descriptive statistics.

Data summary and listings will be presented for subjects who rolled over to 101-99 and sorted by regimen number of the therapy.

#### 7.4. Physical Examination

Physical examination results will be summarized by body system. All results will be listed. Results will be provided on subjects who rolled over to 101-99 only.

## 7.5. Changes From Protocol-Specified Safety Analyses

The protocol specified that data will be summarized by the use or not of concomitant anti-cancer therapy. As anti-cancer therapy is allowed in this study per protocol, a summary will be given for all subjects regardless of taking antitumor treatment or not.

# 8. SOFTWARE

SAS® Software Version 9.2 or higher, SAS Institute Inc., Cary, NC, USA.

# 9. SAP REVISION

| Revision Date (dd month, yyyy) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

### 10. APPENDICES

#### Note:

- "Parent Study +99" (ie, 02+99, 07+99, 08+99, 10+99) indicate combining all subjects in the parent study with data from 101-99
- "99 (parent study)" (ie, 99 (02), 99 (07), 99 (08), 99 (10)) indicate combining only subjects in the parent study who rolled over to 101-99 with data from 101-99
- "99 only" indicate that data presented is from 101-99 only

### **10.1.** Tables

| Table | 1.1.1 | Subject Disposition - 02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 1.1.1.1 | Subject Disposition - 02+99 -CLL | ITT Analysis Set |
| Table | 1.1.1.2 | Subject Disposition - 02+99 -iNHL | ITT Analysis Set |
| Table | 1.1.1.3 | Subject Disposition - 02+99 -MCL | ITT Analysis Set |
| Table | 1.1.1.4 | Subject Disposition - 02+99 -FL | ITT Analysis Set |
| Table | 1.1.1.5 | Subject Disposition - 02+99 -SLL | ITT Analysis Set |
| Table | 1.1.1.6 | Subject Disposition - 02+99 -LPL/WM | ITT Analysis Set |
| Table | 1.1.1.7 | Subject Disposition - 02+99 -MZL | ITT Analysis Set |
| Table | 1.1.2 | Subject Disposition - 07+99 | ITT Analysis Set |
| Table | 1.1.2.1 | Subject Disposition - 07+99- CLL | ITT Analysis Set |
| Table | 1.1.2.2 | Subject Disposition - 07+99- iNHL | ITT Analysis Set |
| Table | 1.1.2.3 | Subject Disposition - 07+99- MCL | ITT Analysis Set |
| Table | 1.1.3 | Subject Disposition -08+99-CLL | ITT Analysis Set |
| Table | 1.1.4 | Subject Disposition - 10+99-iNHL | ITT Analysis Set |
| Table | 1.2.1 | Demographics and Baseline Characteristics -99 (02) | ITT Analysis Set |
| Table | 1.2.1.1 | Demographics and Baseline Characteristics -99 (02) - CLL | ITT Analysis Set |
| Table | 1.2.1.2 | Demographics and Baseline Characteristics - 99 (02)- iNHL | ITT Analysis Set |
| Table | 1.2.1.3 | Demographics and Baseline Characteristics - 99 (02)- MCL | ITT Analysis Set |
| Table | 1.2.1.4 | Demographics and Baseline Characteristics - 99 (02)- FL | ITT Analysis Set |
| Table | 1.2.1.5 | Demographics and Baseline Characteristics - 99 (02)- SLL | ITT Analysis Set |
| Table | 1.2.1.6 | Demographics and Baseline Characteristics - 99 (02)- LPL/WM | ITT Analysis Set |

| Table | 1.2.1.7 | Demographics and Baseline Characteristics - 99 (02)- MZL | ITT Analysis Set |
|---|---|---|---|
| Table | 1.2.2 | Demographics and Baseline Characteristics -99 (07) | ITT Analysis Set |
| Table | 1.2.2.1 | Demographics and Baseline Characteristics -99 (07) - CLL | ITT Analysis Set |
| Table | 1.2.2.2 | Demographics and Baseline Characteristics - 99 (07)- iNHL | ITT Analysis Set |
| Table | 1.2.2.3 | Demographics and Baseline Characteristics - 99 (07)- MCL | ITT Analysis Set |
| Table | 1.2.3 | Demographics and Baseline Characteristics -99 (08)-CLL | ITT Analysis Set |
| Table | 1.2.4 | Demographics and Baseline Characteristics -99 (10)-iNHL | ITT Analysis Set |
| Table | 1.3.1.1 | Disease History -99 (02) - CLL | ITT Analysis Set |
| Table | 1.3.1.2 | Disease History - 99 (02)- iNHL | ITT Analysis Set |
| Table | 1.3.1.3 | Disease History - 99 (02)- MCL | ITT Analysis Set |
| Table | 1.3.1.4 | Disease History - 99 (02)- FL | ITT Analysis Set |
| Table | 1.3.1.5 | Disease History - 99 (02)- SLL | ITT Analysis Set |
| Table | 1.3.1.6 | Disease History - 99 (02)- LPL/WM | ITT Analysis Set |
| Table | 1.3.1.7 | Disease History - 99 (02)- MZL | ITT Analysis Set |
| Table | 1.3.2.1 | Disease History -99 (07) - CLL | ITT Analysis Set |
| Table | 1.3.2.2 | Disease History - 99 (07)- iNHL | ITT Analysis Set |
| Table | 1.3.2.3 | Disease History - 99 (07)- MCL | ITT Analysis Set |
| Table | 1.3.3 | Disease History -99 (08)-CLL | ITT Analysis Set |
| Table | 1.3.4 | Disease History -99 (10)-iNHL | ITT Analysis Set |
| Table | 1.4.1 | Medical History -99 (02) | ITT Analysis Set |
| Table | 1.4.1.1 | Medical History -99 (02) - CLL | ITT Analysis Set |
| Table | 1.4.1.4 | Medical History - 99 (02)- iNHL | ITT Analysis Set |
| Table | 1.4.1.4 | Medical History - 99 (02)- MCL | ITT Analysis Set |
| Table | 1.4.1.4 | Medical History - 99 (02)- FL | ITT Analysis Set |
| Table | 1.4.1.5 | Medical History - 99 (02)- SLL | ITT Analysis Set |
| Table | 1.4.1.6 | Medical History - 99 (02)- LPL/WM | ITT Analysis Set |
| Table | 1.4.1.7 | Medical History - 99 (02)- MZL | ITT Analysis Set |
| Table | 1.4.2 | Medical History -99 (07) | ITT Analysis Set |
| Table | 1.4.2.1 | Medical History -99 (07) - CLL | ITT Analysis Set |
| Table | 1.4.2.2 | Medical History - 99 (07)- iNHL | ITT Analysis Set |
| Table | 1.4.2.3 | Medical History - 99 (07)- MCL | ITT Analysis Set |
| Table | 1.4.3 | Medical History -99 (08)-CLL | ITT Analysis Set |
| Table | 1.4.4 | Medical History -99 (10)-iNHL | ITT Analysis Set |

| Table | 1.5.1 | Physical Examination -99 (02) | ITT Analysis Set |
|-------|---------|----------------------------------------|------------------|
| Table | 1.5.1.1 | Physical Examination -99 (02) - CLL | ITT Analysis Set |
| Table | 1.5.1.5 | Physical Examination - 99 (02)- iNHL | ITT Analysis Set |
| Table | 1.5.1.5 | Physical Examination - 99 (02)- MCL | ITT Analysis Set |
| Table | 1.5.1.5 | Physical Examination - 99 (02)- FL | ITT Analysis Set |
| Table | 1.5.1.5 | Physical Examination - 99 (02)- SLL | ITT Analysis Set |
| Table | 1.5.1.6 | Physical Examination - 99 (02)- LPL/WM | ITT Analysis Set |
| Table | 1.5.1.7 | Physical Examination - 99 (02)- MZL | ITT Analysis Set |
| Table | 1.5.2 | Physical Examination -99 (07) | ITT Analysis Set |
| Table | 1.5.2.1 | Physical Examination -99 (07) - CLL | ITT Analysis Set |
| Table | 1.5.2.2 | Physical Examination - 99 (07)- iNHL | ITT Analysis Set |
| Table | 1.5.2.3 | Physical Examination - 99 (07)- MCL | ITT Analysis Set |
| Table | 1.5.3 | Physical Examination -99 (08)-CLL | ITT Analysis Set |
| Table | 1.5.4 | Physical Examination -99 (10)-iNHL | ITT Analysis Set |
| Table | 1.6.1 | Prior Therapy -99 (02) | ITT Analysis Set |
| Table | 1.6.1.1 | Prior Therapy -99 (02) - CLL | ITT Analysis Set |
| Table | 1.6.1.6 | Prior Therapy - 99 (02)- iNHL | ITT Analysis Set |
| Table | 1.6.1.6 | Prior Therapy - 99 (02)- MCL | ITT Analysis Set |
| Table | 1.6.1.6 | Prior Therapy - 99 (02)- FL | ITT Analysis Set |
| Table | 1.6.1.6 | Prior Therapy - 99 (02)- SLL | ITT Analysis Set |
| Table | 1.6.1.6 | Prior Therapy - 99 (02)- LPL/WM | ITT Analysis Set |
| Table | 1.6.1.7 | Prior Therapy - 99 (02)- MZL | ITT Analysis Set |
| Table | 1.6.2 | Prior Therapy -99 (07) | ITT Analysis Set |
| Table | 1.6.2.1 | Prior Therapy -99 (07) - CLL | ITT Analysis Set |
| Table | 1.6.2.2 | Prior Therapy - 99 (07)- iNHL | ITT Analysis Set |
| Table | 1.6.2.3 | Prior Therapy - 99 (07)- MCL | ITT Analysis Set |
| Table | 1.6.4 | Prior Therapy -99 (10)-iNHL | ITT Analysis Set |
| Table | 1.7.1 | Study Drug Exposure - 02+99 | ITT Analysis Set |
| Table | 1.7.1.1 | Study Drug Exposure - 02+99 -CLL | ITT Analysis Set |
| Table | 1.7.1.2 | Study Drug Exposure - 02+99 -iNHL | ITT Analysis Set |
| Table | 1.7.1.7 | Study Drug Exposure - 02+99 -MCL | ITT Analysis Set |
| Table | 1.7.1.4 | Study Drug Exposure - 02+99 -FL | ITT Analysis Set |
| Table | 1.7.1.5 | Study Drug Exposure - 02+99 -SLL | ITT Analysis Set |
| | | | • |

| Table | 1.7.1.6 | Study Drug Exposure - 02+99 -LPL/WM | ITT Analysis Set |
|---|---|---|---|
| Table | 1.7.1.7 | Study Drug Exposure - 02+99 -MZL | ITT Analysis Set |
| Table | 1.7.2 | Study Drug Exposure - 07+99 | ITT Analysis Set |
| Table | 1.7.2.1 | Study Drug Exposure - 07+99 - CLL | ITT Analysis Set |
| Table | 1.7.2.2 | Study Drug Exposure - 07+99 - iNHL | ITT Analysis Set |
| Table | 1.7.2.3 | Study Drug Exposure - 07+99 - MCL | ITT Analysis Set |
| Table | 1.7.3 | Study Drug Exposure - 08+99 - CLL | ITT Analysis Set |
| Table | 1.7.4 | Study Drug Exposure – 10+99 - iNHL | ITT Analysis Set |
| Table | 2.1.1 | Clinical Response Rate - 02+99 | ITT Analysis Set |
| Table | 2.1.1.1 | Clinical Response Rate - 02+99 -CLL | ITT Analysis Set |
| Table | 2.1.1.2 | Clinical Response Rate - 02+99 -iNHL | ITT Analysis Set |
| Table | 2.1.1.3 | Clinical Response Rate - 02+99 -MCL | ITT Analysis Set |
| Table | 2.1.1.4 | Clinical Response Rate - 02+99 -FL | ITT Analysis Set |
| Table | 2.1.1.5 | Clinical Response Rate - 02+99 -SLL | ITT Analysis Set |
| Table | 2.1.1.6 | Clinical Response Rate - 02+99 -LPL/WM | ITT Analysis Set |
| Table | 2.1.1.7 | Clinical Response Rate - 02+99 -MZL | ITT Analysis Set |
| Table | 2.1.2 | Clinical Response Rate - 07+99 (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.1.2.1 | Clinical Response Rate - 07+99 – CLL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.1.2.2 | Clinical Response Rate - 07+99 – iNHL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.1.3 | Clinical Response Rate - 08+99 - CLL | ITT Analysis Set |
| Table | 2.2.1 | Progression Free Survival - 02+99 | ITT Analysis Set |
| Table | 2.2.1.1 | Progression Free Survival - 02+99 -CLL | ITT Analysis Set |
| Table | 2.2.1.2 | Progression Free Survival - 02+99 -iNHL | ITT Analysis Set |
| Table | 2.2.1.3 | Progression Free Survival - 02+99 -MCL | ITT Analysis Set |
| Table | 2.2.1.4 | Progression Free Survival - 02+99 -FL | ITT Analysis Set |
| Table | 2.2.1.5 | Progression Free Survival - 02+99 -SLL | ITT Analysis Set |
| Table | 2.2.1.6 | Progression Free Survival - 02+99 -LPL/WM | ITT Analysis Set |
| Table | 2.2.1.7 | Progression Free Survival - 02+99 -MZL | ITT Analysis Set |
| Table | 2.2.2 | Progression Free Survival - 07+99 (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.2.2.1 | Progression Free Survival - 07+99 – CLL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.2.2.2 | Progression Free Survival - 07+99 – iNHL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.2.3 | Progression Free Survival - 08+99 - CLL | ITT Analysis Set |
| Table | 2.3.1 | Duration of Response - 02+99 | ITT Analysis Set |
| | • | | |

| Table | 2.3.1.1 | Duration of Response - 02+99 -CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 2.3.1.2 | Duration of Response - 02+99 -iNHL | ITT Analysis Set |
| Table | 2.3.1.3 | Duration of Response - 02+99 -MCL | ITT Analysis Set |
| Table | 2.3.1.4 | Duration of Response - 02+99 -FL | ITT Analysis Set |
| Table | 2.3.1.5 | Duration of Response - 02+99 -SLL | ITT Analysis Set |
| Table | 2.3.1.6 | Duration of Response - 02+99 -LPL/WM | ITT Analysis Set |
| Table | 2.3.1.7 | Duration of Response - 02+99 -MZL | ITT Analysis Set |
| Table | 2.3.2 | Duration of Response - 07+99 (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.3.2.1 | Duration of Response - 07+99 – CLL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.3.2.2 | Duration of Response - 07+99 – iNHL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.3.3 | Duration of Response - 08+99 - CLL | ITT Analysis Set |
| Table | 2.4.1 | Time to Response -02+99 | ITT Analysis Set |
| Table | 2.4.1.1 | Time to Response -02+99 - CLL | ITT Analysis Set |
| Table | 2.4.1.2 | Time to Response -02+99 - iNHL | ITT Analysis Set |
| Table | 2.4.1.3 | Time to Response -02+99 - MCL | ITT Analysis Set |
| Table | 2.4.1.4 | Time to Response -02+99 - FL | ITT Analysis Set |
| Table | 2.4.1.5 | Time to Response -02+99 - SLL | ITT Analysis Set |
| Table | 2.4.1.6 | Time to Response -02+99 - LPL/WM | ITT Analysis Set |
| Table | 2.4.1.7 | Time to Response -02+99 - MZL | ITT Analysis Set |
| Table | 2.4.2 | Time to Response -07+99 (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.4.2.1 | Time to Response - 07+99 – CLL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.4.2.2 | Time to Response - 07+99 – iNHL (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.4.3 | Time to Response - 08+99 - CLL | ITT Analysis Set |
| Table | 2.5.1 | Progression Free Survival - 02+99 (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.1 | Progression Free Survival - 02+99 -CLL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.2 | Progression Free Survival - 02+99 –iNHL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.3 | Progression Free Survival - 02+99 –MCL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.4 | Progression Free Survival - 02+99 -FL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.5 | Progression Free Survival - 02+99 -SLL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.6 | Progression Free Survival - 02+99 -LPL/WM (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.5.1.7 | Progression Free Survival - 02+99 -MZL (Sensitivity Analysis) | ITT Analysis Set |

| Table | 2.5.2 | Progression Free Survival - 07+99 (Sensitivity Analysis) (cohort 1 to 4) | ITT Analysis Set |
|---|---|---|---|
| Table | 2.5.2.1 | Progression Free Survival - 07+99 – CLL (Sensitivity Analysis) (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.5.2.2 | Progression Free Survival - 07+99 – iNHL (Sensitivity Analysis) (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.5.3 | Progression Free Survival - 08+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1 | Duration of Response - 02+99 (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.1 | Duration of Response - 02+99 –CLL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.2 | Duration of Response - 02+99 –iNHL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.3 | Duration of Response - 02+99 –MCL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.4 | Duration of Response - 02+99 -FL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.5 | Duration of Response - 02+99 -SLL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.6 | Duration of Response - 02+99 -LPL/WM (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.1.7 | Duration of Response - 02+99 -MZL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 2.6.2 | Duration of Response - 07+99 (Sensitivity Analysis) (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.6.2.1 | Duration of Response - 07+99 – CLL (Sensitivity Analysis) (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.6.2.2 | Duration of Response - 07+99 – iNHL (Sensitivity Analysis) (cohort 1 to 4) | ITT Analysis Set |
| Table | 2.6.3 | Duration of Response - 08+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Table | 3.1.1 | Overview of Treatment-Emergent Adverse Events – 02+99 | ITT Analysis Set |
| Table | 3.1.1.1 | Overview of Treatment-Emergent Adverse Events – 02+99 – CLL | ITT Analysis Set |
| Table | 3.1.1.2 | Overview of Treatment-Emergent Adverse Events – 02+99 - iNHL | ITT Analysis Set |
| Table | 3.1.1.3 | Overview of Treatment-Emergent Adverse Events – 02+99 - MCL | ITT Analysis Set |
| Table | 3.1.1.4 | Overview of Treatment-Emergent Adverse Events – 02+99 - FL | ITT Analysis Set |
| Table | 3.1.1.5 | Overview of Treatment-Emergent Adverse Events – 02+99 - SLL | ITT Analysis Set |
| Table | 3.1.1.6 | Overview of Treatment-Emergent Adverse Events – 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.1.1.7 | Overview of Treatment-Emergent Adverse Events – 02+99 - MZL | ITT Analysis Set |
| Table | 3.1.2 | Overview of Treatment-Emergent Adverse Events – 07+99 | ITT Analysis Set |

| Table | 3.1.2.1 | Overview of Treatment-Emergent Adverse Events – 07+99 – CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.1.2,2 | Overview of Treatment-Emergent Adverse Events – 07+99 – iNHL | ITT Analysis Set |
| Table | 3.1.2.3 | Overview of Treatment-Emergent Adverse Events – 07+99 – MCL | ITT Analysis Set |
| Table | 3.1.3 | Overview of Treatment-Emergent Adverse Events – 08+99 – CLL | ITT Analysis Set |
| Table | 3.1.4 | Overview of Treatment-Emergent Adverse Events – 10+99 – iNHL | ITT Analysis Set |
| Table | 3.2.1 | Overview of Treatment-Emergent Adverse Events – 99 (02) | ITT Analysis Set |
| Table | 3.2.1.1 | Overview of Treatment-Emergent Adverse Events – 99 (02) – CLL | ITT Analysis Set |
| Table | 3.2.1.2 | Overview of Treatment-Emergent Adverse Events – 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.2.1.3 | Overview of Treatment-Emergent Adverse Events – 99 (02) - MCL | ITT Analysis Set |
| Table | 3.2.1.4 | Overview of Treatment-Emergent Adverse Events – 99 (02) - FL | ITT Analysis Set |
| Table | 3.2.1.5 | Overview of Treatment-Emergent Adverse Events – 99 (02) - SLL | ITT Analysis Set |
| Table | 3.2.1.6 | Overview of Treatment-Emergent Adverse Events – 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.2.1.7 | Overview of Treatment-Emergent Adverse Events – 99 (02) - MZL | ITT Analysis Set |
| Table | 3.2.2 | Overview of Treatment-Emergent Adverse Events – 99 (07) | ITT Analysis Set |
| Table | 3.2.2.1 | Overview of Treatment-Emergent Adverse Events – 99 (07) – CLL | ITT Analysis Set |
| Table | 3.2.2,2 | Overview of Treatment-Emergent Adverse Events – 99 (07) – iNHL | ITT Analysis Set |
| Table | 3.2.2.3 | Overview of Treatment-Emergent Adverse Events – 99 (07) – MCL | ITT Analysis Set |
| Table | 3.2.3 | Overview of Treatment-Emergent Adverse Events – 99 (08) – CLL | ITT Analysis Set |
| Table | 3.2.4 | Overview of Treatment-Emergent Adverse Events – 99 (10) – iNHL | ITT Analysis Set |
| Table | 3.3.1 | Overview of Treatment-Emergent Adverse Events – 99 only (02) | ITT Analysis Set |
| Table | 3.3.1.1 | Overview of Treatment-Emergent Adverse Events – 99 only (02) – CLL | ITT Analysis Set |
| Table | 3.3.1.2 | Overview of Treatment-Emergent Adverse Events – 99 only (02) - iNHL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.3.1.3 | Overview of Treatment-Emergent Adverse Events – 99 only (02) - MCL | ITT Analysis Set |
| Table | 3.3.1.4 | Overview of Treatment-Emergent Adverse Events – 99 only (02) - FL | ITT Analysis Set |
| Table | 3.3.1.5 | Overview of Treatment-Emergent Adverse Events – 99 only (02) - SLL | ITT Analysis Set |
| Table | 3.3.1.6 | Overview of Treatment-Emergent Adverse Events – 99 only (02) - LPL/WM | ITT Analysis Set |
| Table | 3.3.1.7 | Overview of Treatment-Emergent Adverse Events – 99 only (02) - MZL | ITT Analysis Set |
| Table | 3.3.2 | Overview of Treatment-Emergent Adverse Events – 99 only (07) | ITT Analysis Set |
| Table | 3.3.2.1 | Overview of Treatment-Emergent Adverse Events – 99 only (07) – CLL | ITT Analysis Set |
| Table | 3.3.2,2 | Overview of Treatment-Emergent Adverse Events – 99 only (07) – iNHL | ITT Analysis Set |
| Table | 3.3.2.3 | Overview of Treatment-Emergent Adverse Events – 99 only (07) – MCL | ITT Analysis Set |
| Table | 3.3.3 | Overview of Treatment-Emergent Adverse Events – 99 only (08) – CLL | ITT Analysis Set |
| Table | 3.3.4 | Overview of Treatment-Emergent Adverse Events – 99 only (10) – iNHL | ITT Analysis Set |
| Table | 3.4.1 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -02+99 | ITT Analysis Set |
| Table | 3.4.1.1 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – CLL | ITT Analysis Set |
| Table | 3.4.1.2 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – iNHL | ITT Analysis Set |
| Table | 3.4.1.3 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – MCL | ITT Analysis Set |
| Table | 3.4.1.4 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – FL | ITT Analysis Set |
| Table | 3.4.1.5 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – SLL | ITT Analysis Set |
| Table | 3.4.1.6 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.4.1.7 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-02+99 – MZL | ITT Analysis Set |

| Table | | | |
|---|---|---|---|
| Table | 3.4.2 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -07+99 | ITT Analysis Set |
| Table | 3.4.2.1 | Treatment-Emergent Adverse Events by System Organ Class, High Level Term and Preferred Term -07+99 – CLL | ITT Analysis Set |
| Table | 3.4.2.2 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -07+99 – iNHL | ITT Analysis Set |
| Table | 3.4.2.3 | Treatment-Emergent Adverse Events by System Organ Class, High Level Term and Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.4.3 | Treatment-Emergent Adverse Events by System Organ Class, High Level Term and Preferred Term -08+99 – CLL | ITT Analysis Set |
| Table | 3.4.4 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -10+99 – iNHL | ITT Analysis Set |
| Table | 3.5.1 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -99 (02) | ITT Analysis Set |
| Table | 3.5.1.1 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – CLL | ITT Analysis Set |
| Table | 3.5.1.2 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – iNHL | ITT Analysis Set |
| Table | 3.5.1.3 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – MCL | ITT Analysis Set |
| Table | 3.5.1.4 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – FL | ITT Analysis Set |
| Table | 3.5.1.5 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – SLL | ITT Analysis Set |
| Table | 3.5.1.6 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – LPL/WM | ITT Analysis Set |
| Table | 3.5.1.7 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term-99 (02) – MZL | ITT Analysis Set |
| Table | 3.5.2 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -99 (07) | ITT Analysis Set |
| Table | 3.5.2.1 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.5.2.2 | Treatment-Emergent Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.5.2.3 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.5.3 | Treatment-Emergent Adverse Events by System Organ Class,<br>High Level Term and Preferred Term -99 (08) – CLL | ITT Analysis Set |
| Table | 3.5.4 | Treatment-Emergent Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (10) – iNHL | ITT Analysis Set |

| Table | 3.6.1 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 3.6.1.1 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - CLL | ITT Analysis Set |
| Table | 3.6.1.2 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - iNHL | ITT Analysis Set |
| Table | 3.6.1.3 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - MCL | ITT Analysis Set |
| Table | 3.6.1.4 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - FL | ITT Analysis Set |
| Table | 3.6.1.5 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - SLL | ITT Analysis Set |
| Table | 3.6.1.6 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.6.1.7 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - MZL | ITT Analysis Set |
| Table | 3.6.2 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 | ITT Analysis Set |
| Table | 3.6.2.1 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 - CLL | ITT Analysis Set |
| Table | 3.6.2.2 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 - iNHL | ITT Analysis Set |
| Table | 3.6.2.3 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 - MCL | ITT Analysis Set |
| Table | 3.6.3 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>08+99 - CLL | ITT Analysis Set |
| Table | 3.6.4 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term -<br>10+99 - iNHL | ITT Analysis Set |

| Table | 3.7.1 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.7.1.1 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - CLL | ITT Analysis Set |
| Table | 3.7.1.2 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - iNHL | ITT Analysis Set |
| Table | 3.7.1.3 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - MCL | ITT Analysis Set |
| Table | 3.7.1.4 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - FL | ITT Analysis Set |
| Table | 3.7.1.5 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - SLL | ITT Analysis Set |
| Table | 3.7.1.6 | Treatment-Emergent Adverse Events by Severity and by System Organ Class, High Level Term and Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.7.1.7 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - MZL | ITT Analysis Set |
| Table | 3.7.2 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) | ITT Analysis Set |
| Table | 3.7.2.1 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) - CLL | ITT Analysis Set |
| Table | 3.7.2.2 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) - iNHL | ITT Analysis Set |
| Table | 3.7.2.3 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) - MCL | ITT Analysis Set |
| Table | 3.7.3 | Treatment-Emergent Adverse Events by Severity and by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(08) - CLL | ITT Analysis Set |
| Table | 3.7.4 | Treatment-Emergent Adverse Events by Severity and by System Organ Class, High Level Term and Preferred Term - 99 (10) - iNHL | ITT Analysis Set |

| Table | 3.8.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 3.8.1.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.8.1.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.8.1.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.8.1.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.8.1.5 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.8.1.6 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.8.1.7 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.8.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 07+99 | ITT Analysis Set |
| Table | 3.8.2.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 07+99- CLL | ITT Analysis Set |
| Table | 3.8.2.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 07+99- iNHL | ITT Analysis Set |
| Table | 3.8.2.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 07+99- MCL | ITT Analysis Set |
| Table | 3.8.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 08+99 - CLL | ITT Analysis Set |
| Table | 3.8.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 10+99 - iNHL | ITT Analysis Set |

| Table | 3.9.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.9.1.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - CLL | ITT Analysis Set |
| Table | 3.9.1.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - iNHL | ITT Analysis Set |
| Table | 3.9.1.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - MCL | ITT Analysis Set |
| Table | 3.9.1.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - FL | ITT Analysis Set |
| Table | 3.9.1.5 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - SLL | ITT Analysis Set |
| Table | 3.9.1.6 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - LPL/WM | ITT Analysis Set |
| Table | 3.9.1.7 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - MZL | ITT Analysis Set |
| Table | 3.9.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) | ITT Analysis Set |
| Table | 3.9.2.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) - CLL | ITT Analysis Set |
| Table | 3.9.2.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) - iNHL | ITT Analysis Set |
| Table | 3.9.2.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) - MCL | ITT Analysis Set |
| Table | 3.9.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (08) - CLL | ITT Analysis Set |
| Table | 3.9.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (10) - iNHL | ITT Analysis Set |

| Table | 3.10.1 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 3.10.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – CLL | ITT Analysis Set |
| Table | 3.10.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – iNHL | ITT Analysis Set |
| Table | 3.10.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – MCL | ITT Analysis Set |
| Table | 3.10.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – FL | ITT Analysis Set |
| Table | 3.10.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – SLL | ITT Analysis Set |
| Table | 3.10.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.10.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 02+99 – MZL | ITT Analysis Set |
| Table | 3.10.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 | ITT Analysis Set |
| Table | 3.10.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 07+99 – CLL | ITT Analysis Set |
| Table | 3.10.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 07+99 – iNHL | ITT Analysis Set |
| Table | 3.10.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 07+99 – MCL | ITT Analysis Set |
| Table | 3.10.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -<br>08+99 -CLL | ITT Analysis Set |
| Table | 3.10.4 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term - 10+99-iNHL | ITT Analysis Set |

| Table | 3.11.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.11.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – CLL | ITT Analysis Set |
| Table | 3.11.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – iNHL | ITT Analysis Set |
| Table | 3.11.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – MCL | ITT Analysis Set |
| Table | 3.11.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – FL | ITT Analysis Set |
| Table | 3.11.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – SLL | ITT Analysis Set |
| Table | 3.11.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – LPL/WM | ITT Analysis Set |
| Table | 3.11.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(02) – MZL | ITT Analysis Set |
| Table | 3.11.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(07) | ITT Analysis Set |
| Table | 3.11.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.11.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(07) – iNHL | ITT Analysis Set |
| Table | 3.11.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.11.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(08) -CLL | ITT Analysis Set |
| Table | 3.11.4 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>System Organ Class, High Level Term and Preferred Term -99<br>(10)-iNHL | ITT Analysis Set |

| Table | 3.12.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 3.12.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.12.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.12.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.12.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.12.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.12.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.12.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.12.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.12.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.12.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.12.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.12.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.12.4 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 10+99 - iNHL | ITT Analysis Set |

| Table | 3.13.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.13.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.13.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by System Organ Class, High Level Term and Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.13.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.13.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.13.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.13.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.13.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| Table | 3.13.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) | ITT Analysis Set |
| Table | 3.13.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - CLL | ITT Analysis Set |
| Table | 3.13.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.13.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.13.3 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.13.4 | Treatment-Emergent Adverse Events Related to Idelalisib by<br>Severity and by System Organ Class, High Level Term and<br>Preferred Term - 99 (10) - iNHL | ITT Analysis Set |

| Table | 3.14.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 3.14.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- CLL | ITT Analysis Set |
| Table | 3.14.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- iNHL | ITT Analysis Set |
| Table | 3.14.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- MCL | ITT Analysis Set |
| Table | 3.14.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- FL | ITT Analysis Set |
| Table | 3.14.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- SLL | ITT Analysis Set |
| Table | 3.14.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- LPL/WM | ITT Analysis Set |
| Table | 3.14.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 02+99- MZL | ITT Analysis Set |
| Table | 3.14.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 07+99 | ITT Analysis Set |
| Table | 3.14.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 07+99- CLL | ITT Analysis Set |
| Table | 3.14.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 07+99- iNHL | ITT Analysis Set |
| Table | 3.14.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 07+99- MCL | ITT Analysis Set |
| Table | 3.14.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 08+99 - CLL | ITT Analysis Set |
| Table | 3.14.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term – 10+99 - iNHL | ITT Analysis Set |

| Table | 3.15.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.15.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - CLL | ITT Analysis Set |
| Table | 3.15.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - iNHL | ITT Analysis Set |
| Table | 3.15.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - MCL | ITT Analysis Set |
| Table | 3.15.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - FL | ITT Analysis Set |
| Table | 3.15.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - SLL | ITT Analysis Set |
| Table | 3.15.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - LPL/WM | ITT Analysis Set |
| Table | 3.15.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (02) - MZL | ITT Analysis Set |
| Table | 3.15.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) | ITT Analysis Set |
| Table | 3.15.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) - CLL | ITT Analysis Set |
| Table | 3.15.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) - iNHL | ITT Analysis Set |
| Table | 3.15.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (07) - MCL | ITT Analysis Set |
| Table | 3.15.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (08) - CLL | ITT Analysis Set |
| Table | 3.15.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by System Organ Class, High Level Term and Preferred Term - 99 only (10) - iNHL | ITT Analysis Set |

| | | _ | |
|---|---|---|---|
| Table | 3.16.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 | ITT Analysis Set |
| Table | 3.16.1.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – CLL | ITT Analysis Set |
| Table | 3.16.1.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – iNHL | ITT Analysis Set |
| Table | 3.16.1.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – MCL | ITT Analysis Set |
| Table | 3.16.1.4 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – FL | ITT Analysis Set |
| Table | 3.16.1.5 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – SLL | ITT Analysis Set |
| Table | 3.16.1.6 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.16.1.7 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -02+99 – MZL | ITT Analysis Set |
| Table | 3.16.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -07+99 | ITT Analysis Set |
| Table | 3.16.2.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -07+99 – CLL | ITT Analysis Set |
| Table | 3.16.2.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -07+99 – iNHL | ITT Analysis Set |
| Table | 3.16.2.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.16.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -08+99 – CLL | ITT Analysis Set |
| Table | 3.16.4 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -10+99 – iNHL | ITT Analysis Set |
| Table | 3.17.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (02) | ITT Analysis Set |
| Table | 3.17.1.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (02) – CLL | ITT Analysis Set |
| Table | 3.17.1.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (02) – iNHL | ITT Analysis Set |
| Table | 3.17.1.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (02) – MCL | ITT Analysis Set |
| Table | 3.17.1.4 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (02) – FL | ITT Analysis Set |
| Table | 3.17.1.5 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (02) – SLL | ITT Analysis Set |

| Table | 3.17.1.6 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 (02) –<br>LPL/WM | ITT Analysis Set |
|---|---|---|---|
| Table | 3.17.1.7 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 (02) – MZL | ITT Analysis Set |
| Table | 3.17.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (07) | ITT Analysis Set |
| Table | 3.17.2.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.17.2.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.17.2.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.17.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (08) – CLL | ITT Analysis Set |
| Table | 3.17.4 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 (10) – iNHL | ITT Analysis Set |
| Table | 3.18.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (02) | ITT Analysis Set |
| Table | 3.18.1.1 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 only (02) –<br>CLL | ITT Analysis Set |
| Table | 3.18.1.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (02) – iNHL | ITT Analysis Set |
| Table | 3.18.1.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (02) – MCL | ITT Analysis Set |
| Table | 3.18.1.4 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (02) – FL | ITT Analysis Set |
| Table | 3.18.1.5 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 only (02) –<br>SLL | ITT Analysis Set |
| Table | 3.18.1.6 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 only (02) –<br>LPL/WM | ITT Analysis Set |
| Table | 3.18.1.7 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 only (02) –<br>MZL | ITT Analysis Set |
| Table | 3.18.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (07) | ITT Analysis Set |

| Table | 3.18.2.1 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (07) – CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.18.2.2 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (07) – iNHL | ITT Analysis Set |
| Table | 3.18.2.3 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (07) – MCL | ITT Analysis Set |
| Table | 3.18.3 | Treatment-Emergent Serious Adverse Events by System Organ<br>Class, High Level Term and Preferred Term -99 only (08) –<br>CLL | ITT Analysis Set |
| Table | 3.18.4 | Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term and Preferred Term -99 only (10) – iNHL | ITT Analysis Set |
| Table | 3.19.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 | ITT Analysis Set |
| Table | 3.19.1.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – CLL | ITT Analysis Set |
| Table | 3.19.1.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – iNHL | ITT Analysis Set |
| Table | 3.19.1.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – MCL | ITT Analysis Set |
| Table | 3.19.1.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – FL | ITT Analysis Set |
| Table | 3.19.1.5 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – SLL | ITT Analysis Set |
| Table | 3.19.1.6 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.19.1.7 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -02+99 – MZL | ITT Analysis Set |
| Table | 3.19.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -07+99 | ITT Analysis Set |

| Table | 3.19.2.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -07+99 – CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.19.2.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -07+99 – iNHL | ITT Analysis Set |
| Table | 3.19.2.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.19.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -08+99 – CLL | ITT Analysis Set |
| Table | 3.19.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -10+99 – iNHL | ITT Analysis Set |
| Table | 3.20.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) | ITT Analysis Set |
| Table | 3.20.1.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – CLL | ITT Analysis Set |
| Table | 3.20.1.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – iNHL | ITT Analysis Set |
| Table | 3.20.1.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – MCL | ITT Analysis Set |
| Table | 3.20.1.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – FL | ITT Analysis Set |
| Table | 3.20.1.5 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – SLL | ITT Analysis Set |
| Table | 3.20.1.6 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – LPL/WM | ITT Analysis Set |
| Table | 3.20.1.7 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (02) – MZL | ITT Analysis Set |
| Table | 3.20.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (07) | ITT Analysis Set |

| Table | 3.20.2.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (07) – CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.20.2.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.20.2.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.20.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (08) – CLL | ITT Analysis Set |
| Table | 3.20.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by System Organ Class, High Level Term and Preferred Term -99 (10) – iNHL | ITT Analysis Set |
| Table | 3.21.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.21.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.21.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.21.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.21.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.21.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.21.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.21.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.21.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 07+99 | ITT Analysis Set |

| Table | 3.21.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.21.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.21.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.21.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.21.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| Table | 3.22.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) | ITT Analysis Set |
| Table | 3.22.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.22.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.22.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.22.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.22.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.22.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.22.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| Table | 3.22.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) | ITT Analysis Set |

| Table | 3.22.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.22.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.22.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.22.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.22.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by System Organ Class, High Level Term and<br>Preferred Term - 99 (10) - iNHL | ITT Analysis Set |
| Table | 3.23.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.23.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.23.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.23.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.23.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.23.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.23.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.23.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.23.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 07+99 | ITT Analysis Set |

| Table | 3.23.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.23.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.23.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.23.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.23.4 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| Table | 3.24.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) | ITT Analysis Set |
| Table | 3.24.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.24.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.24.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.24.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.24.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.24.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.24.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| Table | 3.24.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) | ITT Analysis Set |

| Table | 3.24.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.24.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.24.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.24.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.24.4 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by System Organ Class, High Level Term and<br>Preferred Term - 99 (10) - iNHL | ITT Analysis Set |
| Table | 3.25.1 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 | ITT Analysis Set |
| Table | 3.25.1.1 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - CLL | ITT Analysis Set |
| Table | 3.25.1.2 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - iNHL | ITT Analysis Set |
| Table | 3.25.1.3 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - MCL | ITT Analysis Set |
| Table | 3.25.1.4 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - FL | ITT Analysis Set |
| Table | 3.25.1.5 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - SLL | ITT Analysis Set |
| Table | 3.25.1.6 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.25.1.7 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>02+99 - MZL | ITT Analysis Set |
| Table | 3.25.2 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 | ITT Analysis Set |

| Table | 3.25.2.1 | Treatment-Emergent Adverse Events Leading to Death by System Organ Class, High Level Term and Preferred Term - 07+99 - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.25.2.2 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 - iNHL | ITT Analysis Set |
| Table | 3.25.2.3 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>07+99 - MCL | ITT Analysis Set |
| Table | 3.25.3 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>08+99 - CLL | ITT Analysis Set |
| Table | 3.25.4 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -<br>10+99 - iNHL | ITT Analysis Set |
| Table | 3.26.1 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) | ITT Analysis Set |
| Table | 3.26.1.1 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - CLL | ITT Analysis Set |
| Table | 3.26.1.2 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - iNHL | ITT Analysis Set |
| Table | 3.26.1.3 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - MCL | ITT Analysis Set |
| Table | 3.26.1.4 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - FL | ITT Analysis Set |
| Table | 3.26.1.5 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - SLL | ITT Analysis Set |
| Table | 3.26.1.6 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - LPL/WM | ITT Analysis Set |
| Table | 3.26.1.7 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(02) - MZL | ITT Analysis Set |
| Table | 3.26.2 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) | ITT Analysis Set |

| Table | 3.26.2.1 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term -99<br>(07) - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.26.2.2 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) - iNHL | ITT Analysis Set |
| Table | 3.26.2.3 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(07) - MCL | ITT Analysis Set |
| Table | 3.26.3 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(08) - CLL | ITT Analysis Set |
| Table | 3.26.4 | Treatment-Emergent Adverse Events Leading to Death by<br>System Organ Class, High Level Term and Preferred Term - 99<br>(10) - iNHL | ITT Analysis Set |
| Table | 3.27.1 | Treatment-Emergent Adverse Events by Preferred Term -02+99 | ITT Analysis Set |
| Table | 3.27.1.1 | Treatment-Emergent Adverse Events by Preferred Term-02+99 – CLL | ITT Analysis Set |
| Table | 3.27.1.2 | Treatment-Emergent Adverse Events by Preferred Term-02+99 – iNHL | ITT Analysis Set |
| Table | 3.27.1.3 | Treatment-Emergent Adverse Events by Preferred Term-02+99 - MCL | ITT Analysis Set |
| Table | 3.27.1.4 | Treatment-Emergent Adverse Events by Preferred Term-02+99 – FL | ITT Analysis Set |
| Table | 3.27.1.5 | Treatment-Emergent Adverse Events by Preferred Term-02+99 - SLL | ITT Analysis Set |
| Table | 3.27.1.6 | Treatment-Emergent Adverse Events by Preferred Term-02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.27.1.7 | Treatment-Emergent Adverse Events by Preferred Term-02+99 - MZL | ITT Analysis Set |
| Table | 3.27.2 | Treatment-Emergent Adverse Events by Preferred Term -07+99 | ITT Analysis Set |
| Table | 3.27.2.1 | Treatment-Emergent Adverse Events by Preferred Term -07+99 – CLL | ITT Analysis Set |
| Table | 3.27.2.2 | Treatment-Emergent Adverse Events by Preferred Term -07+99 – iNHL | ITT Analysis Set |
| Table | 3.27.2.3 | Treatment-Emergent Adverse Events by Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.27.3 | Treatment-Emergent Adverse Events by Preferred Term -08+99 – CLL | ITT Analysis Set |
| Table | 3.27.4 | Treatment-Emergent Adverse Events by Preferred Term -10+99 – iNHL | ITT Analysis Set |

| Table | 3.28.1 | Treatment-Emergent Adverse Events by Preferred Term -99 (02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.28.1.1 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) – CLL | ITT Analysis Set |
| Table | 3.28.1.2 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) – iNHL | ITT Analysis Set |
| Table | 3.28.1.3 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) – MCL | ITT Analysis Set |
| Table | 3.28.1.4 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) – FL | ITT Analysis Set |
| Table | 3.28.1.5 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) – SLL | ITT Analysis Set |
| Table | 3.28.1.6 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.28.1.7 | Treatment-Emergent Adverse Events by Preferred Term-99 (02) – MZL | ITT Analysis Set |
| Table | 3.28.2 | Treatment-Emergent Adverse Events by Preferred Term -99 (07) | ITT Analysis Set |
| Table | 3.28.2.1 | Treatment-Emergent Adverse Events by Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.28.2.2 | Treatment-Emergent Adverse Events by Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.28.2.3 | Treatment-Emergent Adverse Events by Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.28.3 | Treatment-Emergent Adverse Events by Preferred Term -99 (08) – CLL | ITT Analysis Set |
| Table | 3.28.4 | Treatment-Emergent Adverse Events by Preferred Term -99 (10) – iNHL | ITT Analysis Set |
| Table | 3.29.1 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.29.1.1 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.29.1.2 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.29.1.3 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.29.1.4 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.29.1.5 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - SLL | ITT Analysis Set |

| Table | 3.29.1.6 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
|---|---|---|---|
| Table | 3.29.1.7 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.29.2 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.29.2.1 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.29.2.2 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.29.2.3 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.29.3 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.29.4 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| Table | 3.30.1 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) | ITT Analysis Set |
| Table | 3.30.1.1 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.30.1.2 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.30.1.3 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.30.1.4 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.30.1.5 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.30.1.6 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.30.1.7 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| Table | 3.30.2 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (07) | ITT Analysis Set |
| Table | 3.30.2.1 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (07) - CLL | ITT Analysis Set |
| Table | 3.30.2.2 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.30.2.3 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| | | <u> </u> | |

| Table | 3.30.3 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (08) - CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.30.4 | Treatment-Emergent Adverse Events by Severity and by Preferred Term - 99 (10) - iNHL | ITT Analysis Set |
| Table | 3.31.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.31.1.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.31.1.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.31.1.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.31.1.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.31.1.5 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.31.1.6 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.31.1.7 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.31.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.31.2.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.31.2.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.31.2.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.31.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.31.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term – 10+99 - iNHL | ITT Analysis Set |
| Table | 3.32.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) | ITT Analysis Set |
| Table | 3.32.1.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - CLL | ITT Analysis Set |
| Table | 3.32.1.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - iNHL | ITT Analysis Set |
| Table | 3.32.1.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - MCL | ITT Analysis Set |
| | | <u> </u> | |

| Table | 3.32.1.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - FL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.32.1.5 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - SLL | ITT Analysis Set |
| Table | 3.32.1.6 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - LPL/WM | ITT Analysis Set |
| Table | 3.32.1.7 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (02) - MZL | ITT Analysis Set |
| Table | 3.32.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (07) | ITT Analysis Set |
| Table | 3.32.2.1 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (07) - CLL | ITT Analysis Set |
| Table | 3.32.2.2 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (07) - iNHL | ITT Analysis Set |
| Table | 3.32.2.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (07) - MCL | ITT Analysis Set |
| Table | 3.32.3 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (08) - CLL | ITT Analysis Set |
| Table | 3.32.4 | Treatment-Emergent Adverse Events with All Grades and Grade >=3 by Preferred Term - 99 only (10) - iNHL | ITT Analysis Set |
| Table | 3.33.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 | ITT Analysis Set |
| Table | 3.33.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – CLL | ITT Analysis Set |
| Table | 3.33.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – iNHL | ITT Analysis Set |
| Table | 3.33.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – MCL | ITT Analysis Set |
| Table | 3.33.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – FL | ITT Analysis Set |
| Table | 3.33.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – SLL | ITT Analysis Set |
| Table | 3.33.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.33.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -02+99 – MZL | ITT Analysis Set |
| Table | 3.33.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -07+99 | ITT Analysis Set |
| Table | 3.33.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -07+99 – CLL | ITT Analysis Set |
| | | · | |

| Table | 3.33.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -07+99 – iNHL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.33.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.33.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -08+99 -CLL | ITT Analysis Set |
| Table | 3.33.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -10+99-iNHL | ITT Analysis Set |
| Table | 3.34.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) | ITT Analysis Set |
| Table | 3.34.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – CLL | ITT Analysis Set |
| Table | 3.34.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – iNHL | ITT Analysis Set |
| Table | 3.34.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – MCL | ITT Analysis Set |
| Table | 3.34.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – FL | ITT Analysis Set |
| Table | 3.34.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – SLL | ITT Analysis Set |
| Table | 3.34.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – LPL/WM | ITT Analysis Set |
| Table | 3.34.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (02) – MZL | ITT Analysis Set |
| Table | 3.34.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (07) | ITT Analysis Set |
| Table | 3.34.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.34.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.34.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.34.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (08) -CLL | ITT Analysis Set |
| Table | 3.34.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Preferred Term -99 (10)-iNHL | ITT Analysis Set |
| Table | 3.35.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.35.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| | | • | |

| Table | 3.35.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.35.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.35.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.35.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.35.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.35.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.35.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.35.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.35.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.35.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.35.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.35.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| Table | 3.36.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) | ITT Analysis Set |
| Table | 3.36.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.36.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.36.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.36.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.36.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.36.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.36.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| | | | 1 |

| Table | 3.36.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (07) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.36.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (07) - CLL | ITT Analysis Set |
| Table | 3.36.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.36.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.36.3 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.36.4 | Treatment-Emergent Adverse Events Related to Idelalisib by Severity and by Preferred Term - 99 (10) - iNHL | ITT Analysis Set |
| Table | 3.37.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.37.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.37.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.37.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.37.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.37.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.37.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.37.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.37.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.37.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.37.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.37.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.37.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term – 08+99- CLL | ITT Analysis Set |

| Table | 3.37.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term – 10+99- iNHL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.38.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) | ITT Analysis Set |
| Table | 3.38.1.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - CLL | ITT Analysis Set |
| Table | 3.38.1.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - iNHL | ITT Analysis Set |
| Table | 3.38.1.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - MCL | ITT Analysis Set |
| Table | 3.38.1.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - FL | ITT Analysis Set |
| Table | 3.38.1.5 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - SLL | ITT Analysis Set |
| Table | 3.38.1.6 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - LPL/WM | ITT Analysis Set |
| Table | 3.38.1.7 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (02) - MZL | ITT Analysis Set |
| Table | 3.38.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (07) | ITT Analysis Set |
| Table | 3.38.2.1 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (07) - CLL | ITT Analysis Set |
| Table | 3.38.2.2 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (07) - iNHL | ITT Analysis Set |
| Table | 3.38.2.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (07) - MCL | ITT Analysis Set |
| Table | 3.38.3 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (08) - CLL | ITT Analysis Set |
| Table | 3.38.4 | Treatment-Emergent Adverse Events Related to Idelalisib with All Grades and Grade >=3 by Preferred Term - 99 only (10) - iNHL | ITT Analysis Set |

| Table | 3.39.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 | ITT Analysis Set |
|---|---|---|---|
| Table | 3.39.1.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – CLL | ITT Analysis Set |
| Table | 3.39.1.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – iNHL | ITT Analysis Set |
| Table | 3.39.1.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – MCL | ITT Analysis Set |
| Table | 3.39.1.4 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – FL | ITT Analysis Set |
| Table | 3.39.1.5 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – SLL | ITT Analysis Set |
| Table | 3.39.1.6 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.39.1.7 | Treatment-Emergent Serious Adverse Events by Preferred Term -02+99 – MZL | ITT Analysis Set |
| Table | 3.39.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -07+99 | ITT Analysis Set |
| Table | 3.39.2.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -07+99 - CLL | ITT Analysis Set |
| Table | 3.39.2.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -07+99 – iNHL | ITT Analysis Set |
| Table | 3.39.2.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.39.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -08+99 – CLL | ITT Analysis Set |
| Table | 3.39.4 | Treatment-Emergent Serious Adverse Events by Preferred Term -10+99 – iNHL | ITT Analysis Set |
| Table | 3.40.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) | ITT Analysis Set |
| Table | 3.40.1.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – CLL | ITT Analysis Set |
| Table | 3.40.1.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – iNHL | ITT Analysis Set |
| Table | 3.40.1.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – MCL | ITT Analysis Set |
| Table | 3.40.1.4 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – FL | ITT Analysis Set |
| Table | 3.40.1.5 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – SLL | ITT Analysis Set |
| | | | · |

| Table | 3.40.1.6 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – LPL/WM | ITT Analysis Set |
|---|---|---|---|
| Table | 3.40.1.7 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (02) – MZL | ITT Analysis Set |
| Table | 3.40.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (07) | ITT Analysis Set |
| Table | 3.40.2.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.40.2.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.40.2.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.40.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (08) – CLL | ITT Analysis Set |
| Table | 3.40.4 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 (10) – iNHL | ITT Analysis Set |
| Table | 3.41.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) | ITT Analysis Set |
| Table | 3.41.1.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – CLL | ITT Analysis Set |
| Table | 3.41.1.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – iNHL | ITT Analysis Set |
| Table | 3.41.1.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – MCL | ITT Analysis Set |
| Table | 3.41.1.4 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – FL | ITT Analysis Set |
| Table | 3.41.1.5 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – SLL | ITT Analysis Set |
| Table | 3.41.1.6 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – LPL/WM | ITT Analysis Set |
| Table | 3.41.1.7 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (02) – MZL | ITT Analysis Set |
| Table | 3.41.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (07) | ITT Analysis Set |
| Table | 3.41.2.1 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (07) – CLL | ITT Analysis Set |
| Table | 3.41.2.2 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (07) – iNHL | ITT Analysis Set |
| Table | 3.41.2.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (07) – MCL | ITT Analysis Set |
| | • | | |

| Table | 3.41.3 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (08) – CLL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.41.4 | Treatment-Emergent Serious Adverse Events by Preferred Term -99 only (10) – iNHL | ITT Analysis Set |
| Table | 3.42.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 | ITT Analysis Set |
| Table | 3.42.1.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – CLL | ITT Analysis Set |
| Table | 3.42.1.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – iNHL | ITT Analysis Set |
| Table | 3.42.1.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – MCL | ITT Analysis Set |
| Table | 3.42.1.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – FL | ITT Analysis Set |
| Table | 3.42.1.5 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – SLL | ITT Analysis Set |
| Table | 3.42.1.6 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – LPL/WM | ITT Analysis Set |
| Table | 3.42.1.7 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -02+99 – MZL | ITT Analysis Set |
| Table | 3.42.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -07+99 | ITT Analysis Set |
| Table | 3.42.2.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -07+99 – CLL | ITT Analysis Set |
| Table | 3.42.2.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -07+99 – iNHL | ITT Analysis Set |
| Table | 3.42.2.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -07+99 – MCL | ITT Analysis Set |
| Table | 3.42.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -08+99 – CLL | ITT Analysis Set |
| Table | 3.42.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -10+99 – iNHL | ITT Analysis Set |
| Table | 3.43.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) | ITT Analysis Set |
| Table | 3.43.1.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – CLL | ITT Analysis Set |
| Table | 3.43.1.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – iNHL | ITT Analysis Set |
| Table | 3.43.1.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – MCL | ITT Analysis Set |
| | | · | 1 |

| Table | 3.43.1.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – FL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.43.1.5 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – SLL | ITT Analysis Set |
| Table | 3.43.1.6 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – LPL/WM | ITT Analysis Set |
| Table | 3.43.1.7 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (02) – MZL | ITT Analysis Set |
| Table | 3.43.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (07) | ITT Analysis Set |
| Table | 3.43.2.1 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (07) – CLL | ITT Analysis Set |
| Table | 3.43.2.2 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (07) – iNHL | ITT Analysis Set |
| Table | 3.43.2.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (07) – MCL | ITT Analysis Set |
| Table | 3.43.3 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (08) – CLL | ITT Analysis Set |
| Table | 3.43.4 | Treatment-Emergent Serious Adverse Events Related to Idelalisib by Preferred Term -99 (10) – iNHL | ITT Analysis Set |
| Table | 3.44.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose Reduction by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.44.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.44.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.44.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose Reduction by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.44.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.44.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.44.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.44.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.44.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose Reduction by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.44.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose Reduction by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| | • | • | • |

| Table | 3.44.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose Reduction by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.44.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose Reduction by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.44.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.44.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| Table | 3.45.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) | ITT Analysis Set |
| Table | 3.45.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.45.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.45.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.45.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.45.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.45.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.45.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| Table | 3.45.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (07) | ITT Analysis Set |
| Table | 3.45.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (07) - CLL | ITT Analysis Set |
| Table | 3.45.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.45.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.45.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.45.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Dose<br>Reduction by Preferred Term - 99 (10) - iNHL | ITT Analysis Set |
| Table | 3.46.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.46.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| | • | • | |

| Table | 3.46.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
|---|---|---|---|
| Table | 3.46.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.46.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.46.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.46.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.46.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.46.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.46.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.46.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.46.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.46.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.46.4 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| Table | 3.47.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 99 (02) | ITT Analysis Set |
| Table | 3.47.1.1 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.47.1.2 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.47.1.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.47.1.4 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.47.1.5 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.47.1.6 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.47.1.7 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| | | · | 1 |

| Table | 3.47.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 99 (07) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.47.2.1 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 99 (07) - CLL | ITT Analysis Set |
| Table | 3.47.2.2 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.47.2.3 | Treatment-Emergent Adverse Events Leading to Idelalisib Discontinuation by Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.47.3 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.47.4 | Treatment-Emergent Adverse Events Leading to Idelalisib<br>Discontinuation by Preferred Term - 99 (10) - iNHL | ITT Analysis Set |
| Table | 3.48.1 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 | ITT Analysis Set |
| Table | 3.48.1.1 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - CLL | ITT Analysis Set |
| Table | 3.48.1.2 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - iNHL | ITT Analysis Set |
| Table | 3.48.1.3 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - MCL | ITT Analysis Set |
| Table | 3.48.1.4 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - FL | ITT Analysis Set |
| Table | 3.48.1.5 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - SLL | ITT Analysis Set |
| Table | 3.48.1.6 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - LPL/WM | ITT Analysis Set |
| Table | 3.48.1.7 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 02+99 - MZL | ITT Analysis Set |
| Table | 3.48.2 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 07+99 | ITT Analysis Set |
| Table | 3.48.2.1 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 07+99 - CLL | ITT Analysis Set |
| Table | 3.48.2.2 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 07+99 - iNHL | ITT Analysis Set |
| Table | 3.48.2.3 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 07+99 - MCL | ITT Analysis Set |
| Table | 3.48.3 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 08+99 - CLL | ITT Analysis Set |
| Table | 3.48.4 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 10+99 - iNHL | ITT Analysis Set |
| | • | • | |

| Table | 3.49.1 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) | ITT Analysis Set |
|---|---|---|---|
| Table | 3.49.1.1 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - CLL | ITT Analysis Set |
| Table | 3.49.1.2 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - iNHL | ITT Analysis Set |
| Table | 3.49.1.3 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - MCL | ITT Analysis Set |
| Table | 3.49.1.4 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - FL | ITT Analysis Set |
| Table | 3.49.1.5 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - SLL | ITT Analysis Set |
| Table | 3.49.1.6 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - LPL/WM | ITT Analysis Set |
| Table | 3.49.1.7 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (02) - MZL | ITT Analysis Set |
| Table | 3.49.2 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (07) | ITT Analysis Set |
| Table | 3.49.2.1 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (07) - CLL | ITT Analysis Set |
| Table | 3.49.2.2 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (07) - iNHL | ITT Analysis Set |
| Table | 3.49.2.3 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (07) - MCL | ITT Analysis Set |
| Table | 3.49.3 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (08) - CLL | ITT Analysis Set |
| Table | 3.49.4 | Treatment-Emergent Adverse Events Leading to Death by Preferred Term - 99 (10) - iNHL | ITT Analysis Set |

## 10.2. Listings

| Listing | 1.1.1 | Subject Disposition - 02+99 | ITT Analysis Set |
|---------|-------|-----------------------------|------------------|
| Listing | 1.1.2 | Subject Disposition - 07+99 | ITT Analysis Set |
| Listing | 1.1.3 | Subject Disposition - 08+99 | ITT Analysis Set |
| Listing | 1.1.4 | Subject Disposition - 10+99 | ITT Analysis Set |
| Listing | 1.2.1 | Demographics - 99 (02) | ITT Analysis Set |
| Listing | 1.2.2 | Demographics - 99 (07) | ITT Analysis Set |
| Listing | 1.2.3 | Demographics - 99 (08) | ITT Analysis Set |
| Listing | 1.2.4 | Demographics – 99 (10) | ITT Analysis Set |
| Listing | 1.3.1 | Disease History - 99 (02) | ITT Analysis Set |

| Listing | 1.3.2.1 | Disease History - 99 (07) - CLL | ITT Analysis Set |
|---|---|---|---|
| Listing | 1.3.2.2 | Disease History - 99 (07) – iNHL | ITT Analysis Set |
| Listing | 1.3.2.3 | Disease History - 99 (07) - MCL | ITT Analysis Set |
| Listing | 1.3.3 | Disease History - 99 (08) | ITT Analysis Set |
| Listing | 1.3.4 | Disease History – 99 (10) | ITT Analysis Set |
| Listing | 1.4.1 | Medical History - 99 (02) | ITT Analysis Set |
| Listing | 1.4.2 | Medical History - 99 (07) | ITT Analysis Set |
| Listing | 1.4.3 | Medical History - 99 (08) | ITT Analysis Set |
| Listing | 1.4.4 | Medical History – 99 (10) | ITT Analysis Set |
| Listing | 1.5.1 | Physical Examination - 99 (02) | ITT Analysis Set |
| Listing | 1.5.2 | Physical Examination - 99 (07) | ITT Analysis Set |
| Listing | 1.5.3 | Physical Examination - 99 (08) | ITT Analysis Set |
| Listing | 1.5.4 | Physical Examination – 99 (10) | ITT Analysis Set |
| Listing | 1.6.1 | Prior Therapy - 99 (02) | ITT Analysis Set |
| Listing | 1.6.2 | Prior Therapy - 99 (07) | ITT Analysis Set |
| Listing | 1.6.3 | Prior Therapy – 99 (10) | ITT Analysis Set |
| Listing | 1.7.1 | Subject ID in Parent Study and in 101-99 | ITT Analysis Set |
| Listing | 2.1.1 | Investigator's Response Assessment - 02+99 | ITT Analysis Set |
| Listing | 2.1.2 | Investigator's Response Assessment - 07+99 | ITT Analysis Set |
| Listing | 2.1.3 | Investigator's Response Assessment - 08+99 | ITT Analysis Set |
| Listing | 2.2.1 | Progression Free Survival, Time to Response and Duration of Response - 02+99 | ITT Analysis Set |
| Listing | 2.2.2 | Progression Free Survival, Time to Response and Duration of Response - 07+99 | ITT Analysis Set |
| Listing | 2.2.3 | Progression Free Survival, Time to Response and Duration of Response - 08+99 | ITT Analysis Set |
| Listing | 3.1.1 | Adverse Events - 99 only (02) | ITT Analysis Set |
| Listing | 3.1.2 | Adverse Events - 99 only (07) | ITT Analysis Set |
| Listing | 3.1.3 | Adverse Events - 99 only (08) | ITT Analysis Set |
| Listing | 3.1.4 | Adverse Events - 99 only (10) | ITT Analysis Set |
| Listing | 3.2.1 | Adverse Events Leading to Idelalisib Dose Reduction - 99 only (02) | ITT Analysis Set |
| Listing | 3.2.2 | Adverse Events Leading to Idelalisib Dose Reduction - 99 only (07) | ITT Analysis Set |
| Listing | 3.2.3 | Adverse Events Leading to Idelalisib Dose Reduction - 99 only (08) | ITT Analysis Set |

| Listing | 3.2.4 | Adverse Events Leading to Idelalisib Dose Reduction - 99 only (10) | ITT Analysis Set |
|---|---|---|---|
| Listing | 3.3.1 | Adverse Events Leading to Early Study Withdrawal - 99 only (02) | ITT Analysis Set |
| Listing | 3.3.2 | Adverse Events Leading to Early Study Withdrawal - 99 only (07) | ITT Analysis Set |
| Listing | 3.3.3 | Adverse Events Leading to Early Study Withdrawal - 99 only (08) | ITT Analysis Set |
| Listing | 3.3.4 | Adverse Events Leading to Early Study Withdrawal - 99 only (10) | ITT Analysis Set |
| Listing | 3.4.1 | Adverse Events Leading to Death-99 only (02) | ITT Analysis Set |
| Listing | 3.4.2 | Adverse Events Leading to Death-99 only (07) | ITT Analysis Set |
| Listing | 3.4.3 | Adverse Events Leading to Death-99 only (08) | ITT Analysis Set |
| Listing | 3.4.4 | Adverse Events Leading to Death-99 only (10) | ITT Analysis Set |
| Listing | 3.5.1 | Serious Adverse Events - 99 only (02) | ITT Analysis Set |
| Listing | 3.5.2 | Serious Adverse Events - 99 only (07) | ITT Analysis Set |
| Listing | 3.5.3 | Serious Adverse Events - 99 only (08) | ITT Analysis Set |
| Listing | 3.5.4 | Serious Adverse Events - 99 only (10) | ITT Analysis Set |
| Listing | 4.1.1 | Protocol Violation -99 only (02) | ITT Analysis Set |
| Listing | 4.1.2 | Protocol Violation -99 only (07) | ITT Analysis Set |
| Listing | 4.1.3 | Protocol Violation -99 only (08) | ITT Analysis Set |
| Listing | 4.1.4 | Protocol Violation – 99 only (10) | ITT Analysis Set |
| Listing | 5.1.1 | Concomitant Medication 99 only (02) | ITT Analysis Set |
| Listing | 5.1.2 | Concomitant Medication 99 only (07) | ITT Analysis Set |
| Listing | 5.1.3 | Concomitant Medication 99 only (08) | ITT Analysis Set |
| Listing | 5.1.4 | Concomitant Medication 99 only (10) | ITT Analysis Set |

## 10.3. Figures

| Figure | 1.1.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - CLL | ITT Analysis Set |
|---|---|---|---|
| Figure | 1.1.2 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - iNHL | ITT Analysis Set |
| Figure | 1.1.3 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - MCL | ITT Analysis Set |
| Figure | 1.1.8 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - FL | ITT Analysis Set |
| Figure | 1.1.9 | Kaplan-Meier Plot of Progression Free Survival - 02+99 -SLL | ITT Analysis Set |
| Figure | 1.1.10 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - LPL/WM | ITT Analysis Set |

| | T | T | T |
|---|---|---|---|
| Figure | 1.1.11 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - MZL | ITT Analysis Set |
| Figure | 1.2.1 | Kaplan-Meier Plot of Progression Free Survival - 07+99 - CLL | ITT Analysis Set |
| Figure | 1.2.2 | Kaplan-Meier Plot of Progression Free Survival - 07+99 - iNHL | ITT Analysis Set |
| Figure | 1.3.1 | Kaplan-Meier Plot of Progression Free Survival - 08+99 - CLL | ITT Analysis Set |
| Figure | 2.1.1 | Kaplan-Meier Plot of Duration of Response - 02+99 - CLL | ITT Analysis Set |
| Figure | 2.1.2 | Kaplan-Meier Plot of Duration of Response - 02+99 - iNHL | ITT Analysis Set |
| Figure | 2.1.3 | Kaplan-Meier Plot of Duration of Response - 02+99 - MCL | ITT Analysis Set |
| Figure | 2.1.8 | Kaplan-Meier Plot of Duration of Response - 02+99 - FL | ITT Analysis Set |
| Figure | 2.1.9 | Kaplan-Meier Plot of Duration of Response - 02+99 -SLL | ITT Analysis Set |
| Figure | 2.1.10 | Kaplan-Meier Plot of Duration of Response - 02+99 - LPL/WM | ITT Analysis Set |
| Figure | 2.1.11 | Kaplan-Meier Plot of Duration of Response - 02+99 - MZL | ITT Analysis Set |
| Figure | 2.2.1 | Kaplan-Meier Plot of Duration of Response - 07+99 - CLL | ITT Analysis Set |
| Figure | 2.2.2 | Kaplan-Meier Plot of Duration of Response - 07+99 - iNHL | ITT Analysis Set |
| Figure | 2.3.1 | Kaplan-Meier Plot of Duration of Response - 08+99 - CLL | ITT Analysis Set |
| Figure | 1.1.1.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.1.2.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 – iNHL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.1.3.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 – MCL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.1.8.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 – FL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.1.9.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 –SLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.1.10.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 - LPL/WM (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.1.11.1 | Kaplan-Meier Plot of Progression Free Survival - 02+99 – MZL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.2.1.1 | Kaplan-Meier Plot of Progression Free Survival - 07+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.2.2.1 | Kaplan-Meier Plot of Progression Free Survival - 07+99 – iNHL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 1.3.1.1 | Kaplan-Meier Plot of Progression Free Survival - 08+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.1.1.1 | Kaplan-Meier Plot of Duration of Response - 02+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.1.2.1 | Kaplan-Meier Plot of Duration of Response - 02+99 – iNHL (Sensitivity Analysis) | ITT Analysis Set |

| Figure | 2.1.3.1 | Kaplan-Meier Plot of Duration of Response - 02+99 – MCL (Sensitivity Analysis) | ITT Analysis Set |
|---|---|---|---|
| Figure | 2.1.8.1 | Kaplan-Meier Plot of Duration of Response - 02+99 – FL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.1.9.1 | Kaplan-Meier Plot of Duration of Response - 02+99 –SLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.1.10.1 | Kaplan-Meier Plot of Duration of Response - 02+99 - LPL/WM (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.1.11.1 | Kaplan-Meier Plot of Duration of Response - 02+99 – MZL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.2.1.1 | Kaplan-Meier Plot of Duration of Response - 07+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.2.2.1 | Kaplan-Meier Plot of Duration of Response - 07+99 – iNHL (Sensitivity Analysis) | ITT Analysis Set |
| Figure | 2.3.1.1 | Kaplan-Meier Plot of Duration of Response - 08+99 – CLL (Sensitivity Analysis) | ITT Analysis Set |